CLINICAL TRIAL: NCT00353717
Title: Phase II of Combined Treatment of Cetuximab and Paclitaxel in Basal Like Breast Carcinoma
Brief Title: Combined Treatment of Cetuximab and Paclitaxel in Basal Like Breast Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr Hovav Nechushtan, Hadassah Hebrew university medical center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: cpblb1-HMO-CTIL
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-02

CONDITIONS: Breast Neoplasms
Keywords: breast; basal like; carcinoma; metastatic; EGFR
MeSH Terms: conditions — Breast Neoplasms; Carcinoma; Neoplasm Metastasis | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: cetuximab paclitaxel

INTERVENTIONS:
Drug: cetuximab paclitaxel — weekly iv paclitaxel 80 mg/m2 and cetuximab 250 mg /m2
  Other Names: weekly iv paclitaxel 80 mg/m2 and cetuximab 250 mg /m2

SUMMARY:
Basal like breast carcinoma is a Her2, estrogen receptor (ER) progesterone receptor (PR) negative breast cancer. It is notable for the high level of epidermal growth factor receptor (EGFR) expression in this tumor subtype .

Thus the investigators wanted to combine the use of anti EGFR therapy in the form of Erbitux (cetuximab) with the widely used weekly taxol chemotherapy for the treatment of these women. This is a small phase I/II study.

DETAILED DESCRIPTION:
Basal like breast carcinoma is a Her2, ER PR negative breast cancer. It is notable for the high percentage of EGFR expression in this tumor subtype.Weekly taxol (paclitaxel) is widely used in breast cancer patients with metastatic disease. Erbitux (cetuximab) is a monoclonal antibody that shown its ability to enhance activity of chemotherapy in colon carcinoma. Thus we wanted to combine the use of anti EGFR therapy in the form of Erbitux (cetuximab) with the widely used weekly taxol chemotherapy for the treatment of women with basal like breast carcinoma. This is a small phase II study that will hopefully provide initial data as to the general tolerability and response rate of this combination in this disease. Furthermore, pathologic analysis will be used to try and assess relation of response with the presence of immunohistochemical markers such as EGFR expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast carcinoma of the basal like subtype with available biopsy for analysis and ECOG PS of 2 or less

Exclusion Criteria:

* Pregnancy
* BUN, blood creatinine, AST, ALT > X3 of upper limits of normal
* More than previous 2 chemotherapy lines in the metastatic settings or the use of previous inhibitors of EGFR

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-11; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
tumor markers tumor size by ct | two years

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nechushtan, MD/PHD, Principal Investigator — Hadassah Ein Kerem Jerusalem; Tamar Peretz, MD, Principal Investigator — Hadassah Ein Kerem
Locations (1):
- Oncology Department Hadassah Ein Kerem POB 12000, Jerusalem, Israel

REFERENCES:
- [Background] Nielsen TO, Hsu FD, Jensen K, Cheang M, Karaca G, Hu Z, Hernandez-Boussard T, Livasy C, Cowan D, Dressler L, Akslen LA, Ragaz J, Gown AM, Gilks CB, van de Rijn M, Perou CM. Immunohistochemical and clinical characterization of the basal-like subtype of invasive breast carcinoma. Clin Cancer Res. 2004 Aug 15;10(16):5367-74. doi: 10.1158/1078-0432.CCR-04-0220. PMID 15328174